CLINICAL TRIAL: NCT02722317
Title: Intimate Partner Violence: the Intervention for Men Who Batter Women
Brief Title: Intervention for Men Who Batter Women
Status: Completed | Type: Observational
Sponsor: Santa Catarina Federal University (Other)
Responsible Party: Principal Investigator, Anne Caroline Luz Grudtner da Silva, Master, Santa Catarina Federal University
Other Study IDs: SantaCatarinaFU
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Violence

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: psychological support — psychological support was given to men by the service, the researcher didn't interfered in the intervention, just ask questions about it.

SUMMARY:
It was realized a case study in a batterer intervention program, where 86 men accepted to participate. It was used the Centers for Disease Control and Prevention - Follow up questionnaire, adapted to be used in Brazil.

DETAILED DESCRIPTION:
The intimate partner violence is one of the most common forms of violence. Although man is the main author of violence, it is essential include actions to help him in order to produce a more effective result, because it is believed that he is able to recognize and take responsibility for the violence, using different forms of express. However, these actions have difficulties in evaluating its results. These research aims to analyze the relapse of violence after participation in a batterer intervention program. The investigators realized a case study in a batterer intervention program in the city of Brasília, capital of Brazil, 167 men were invited and 86 accepted to participate of the research. It was used the Centers for Disease Control and Prevention - Follow up questionnaire, adapted to be used in Brazil. All the participants answered the same questionnaire, and the participant exclusion criteria was less or more than 3 months of participation at the program or committed other types of violence. The participants were recruited and interviewed by the investigators, during the year of 2015 (from March until December), in the Center for Assistance to Family and perpetrators of Domestic Violence (NAFAVD). The participants answered questions about socioeconomic characteristics, the relapse of violence, use of drugs, and about the batterer program. The benefit of participate of the study is help to improve the programs to prevent intimate partner violence, and public policy about this issue, and the risk is to remember something that happened during the interview, so the participants could stop the participate when they want.

ELIGIBILITY:
Inclusion Criteria:

* men who participate of the program for 3 months, because committed intimate partner violence

Exclusion Criteria:

* men with less or more than 3 months of participation at the program, or committed other types of violence

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men follow by a batterer intervention program in the city of Brasília, capital of Brazil
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
the relapse of violence after participation in a batterer intervention program | 3 months
  if they committed violence after 3 months, using a questionnaire - yes (physical, sexual or psychology violence)/no/no contact with women

CONTACTS AND LOCATIONS:
Overall Officials: Elza Coelho, Doctor, Study Chair — Santa Catarina Federal University
Locations (1):
- NAFAVD - Núcleo de Atendimento a Núcleo de Atendimento à Família e aos autores de violência Doméstica (Center for Assistance to Family and perpetrators of Domestic violence), Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No